CLINICAL TRIAL: NCT04627584
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled Phase 2 Clinical Trial of MW33 Injection to Evaluate the Efficacy and Safety in Patients With Mild or Moderate COVID-19
Brief Title: A Phase 2 Clinical Trial of MW33 Injection in Patients With COVID-19
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mabwell (Shanghai) Bioscience Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MW33-2020-CP201
Record Dates: First submitted 2020-11-12; First posted 2020-11-13 (Actual); Last update posted 2021-02-26 (Actual); Status verified 2021-02

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- MW33 injection-1200mg (Active Comparator)
  Interventions: Combination Product: MW33 injection
- MW33 injection-2400mg (Active Comparator)
  Interventions: Combination Product: MW33 injection
- Placebo (Placebo Comparator)
  Interventions: Combination Product: MW33 injection placebo

INTERVENTIONS:
Combination Product: MW33 injection — a recombinant fully human antibody to coronavirus
  Arms: MW33 injection-1200mg; MW33 injection-2400mg
Combination Product: MW33 injection placebo — Placebo
  Arms: Placebo

SUMMARY:
This study is designed as a multicenter, randomized, double-blind, placebo-controlled clinical trial to evaluate the clinical efficacy and safety of MW33 injection in patients with mild or moderate COVID-19, and to evaluate its pharmacokinetic profile and immunogenicity.

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed with mild or moderate COVID-19 (as per the Diagnosis and Treatment Protocol for Novel Coronavirus Pneumonia (Trial, 8th edition), China, or Clinical Management of COVID-19, WHO);
2. Has at least one COVID-19 symptom, e.g., fever, cough, shortness of breath, sore throat, headache, muscle ache, and other respiratory or gastrointestinal symptoms, and has the symptom for ≤ 7 days prior to randomization;
3. The SARS-CoV-2 nasopharyngeal nucleic acid is tested to be positive (RT-PCR), IgM (-)/IgG (-) or IgM (+)/IgG (-) within 3 days before randomization;
4. Male or female subjects aged 18 to 80 years (including 18 and 80 years);
5. Subjects do not have a pregnancy plan, voluntarily take effective contraceptive measures during the screening period and the next 6 months, and have no sperm and egg donation plans, and voluntarily take non-pharmaceutical contraception measures during the trial period;
6. Subjects voluntarily sign the informed consent form (ICF) based on sufficient knowledge of the nature, purpose, and procedures of the study, and shall be willing to comply with the study regulations.

Exclusion Criteria:

1. A subject who was diagnosed with severe or critical COVID-19 (as per the Diagnosis and Treatment Protocol for Novel Coronavirus Pneumonia (Trial, 8th edition), China, or Clinical Management of COVID-19, WHO);
2. Abnormal important organ function indicators, which meet the following conditions:

   ① Liver function: serum aspartate aminotransferase (AST) and serum alanine aminotransferase (ALT) > 5.0 × upper limit of normal (ULN);

   ② Renal function: patients treated with dialysis or eGFR< 60 mL/min.

   ③ Cardiac function: patients with results of 12-lead ECG suggesting conduction block or acute myocardial infarction requiring urgent management;
3. Suspected or diagnosed with serious bacterial, fungal, viral, or other infection (except SARS-CoV-2 infection). In the opinion of the investigator, the conditions will prevent a subject from completing the study or impact interpretation of the study results;
4. Currently suffering from serious systemic diseases or mental disorders, and ineligible to participate in the study judged by the investigator;
5. A history of severe trauma, fracture, or surgery within 4 weeks prior to screening, or possibility of requiring a major surgery during the study;
6. Participated in clinical trials of SARS-CoV-2 vaccine or SARS-CoV-2 monoclonal antibody;
7. Received or being receiving the convalescent plasma from patients recovered from COVID-19;
8. Prior or current use of antiviral drugs for treatment of COVID-19, including Remdesivir, Tocilizumab, Interferon, Ribavirin, Abidol, Lopinavir, and Ritonavir, etc.
9. Currently enrolled into clinical studies with other drugs or devices; the time to start of this study from the end of previous participation in other drug clinical studies is less than 30 days, or within 5 half-lives, or within the biological effect period of the drug (whichever is longer);
10. Those who are known to be allergic to any component of the investigational product; or those who have a history of allergies and judged by the investigator to be ineligible for enrollment;
11. Females who are pregnant or lactating;
12. Any conditions that are not suitable for enrollment judged by the investigator.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2020-12-29 (Actual); Primary Completion 2021-05 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
SARS-CoV-2 viral load | 7 Days
  Change in time-weighted SARS-CoV-2 viral load in nasopharyngeal swabs from baseline to day 7

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Public Health Clinical Center, Shanghai, China

REFERENCES:
- [Derived] Kreuzberger N, Hirsch C, Chai KL, Tomlinson E, Khosravi Z, Popp M, Neidhardt M, Piechotta V, Salomon S, Valk SJ, Monsef I, Schmaderer C, Wood EM, So-Osman C, Roberts DJ, McQuilten Z, Estcourt LJ, Skoetz N. SARS-CoV-2-neutralising monoclonal antibodies for treatment of COVID-19. Cochrane Database Syst Rev. 2021 Sep 2;9(9):CD013825. doi: 10.1002/14651858.CD013825.pub2. PMID 34473343
- [Derived] Meng X, Wang P, Xiong Y, Wu Y, Lin X, Lu S, Li R, Zhao B, Liu J, Zeng S, Zeng L, Wu Y, Lu Y, Zhang J, Liu D, Wang S, Lu H. Safety, tolerability, pharmacokinetic characteristics, and immunogenicity of MW33: a Phase 1 clinical study of the SARS-CoV-2 RBD-targeting monoclonal antibody. Emerg Microbes Infect. 2021 Dec;10(1):1638-1648. doi: 10.1080/22221751.2021.1960900. PMID 34346827